CLINICAL TRIAL: NCT04561895
Title: Genetic Variations in Adipokine to Improve Risk Prediction for NAFLD and Its Progression to NASH in Egyptian Patients
Brief Title: Adipokine Genetic Variations in predictingNAFLD Progression to NASH in Egyptian Patients
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Elsahel teaching hospital (Unknown)
Responsible Party: Principal Investigator, Dalia K. Zaafar, lecturer of pharmacology, Cairo University
Other Study IDs: LC ElSahel
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: NAFLD; NASH - Nonalcoholic Steatohepatitis
Keywords: Egyptian population; NAFLD; NASH; DNA extraction; liver enzymes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group: healthy volunteers with absence of NAFLD
  Interventions: Genetic: DNA extraction
- test group: patients with confirmed NAFLD diagnosis
  Interventions: Genetic: DNA extraction

INTERVENTIONS:
Genetic: DNA extraction — investigation of DNA polymorphism in patients suffering from NAFLD

SUMMARY:
Due to the limited data concerning Egyptian population. authors aimed to investigate the differentadipokine gene polymorphism related to non alcoholic fatty liver disease incidence, prognosis and progression to steotosis and also to find different related factors including obesitu, diabetes and liver enzymes level

ELIGIBILITY:
Inclusion Criteria:

Egyptian patients confirmed NAFLD diagnosis diabetic

-

Exclusion Criteria:

* Pregnancy and lactation, history of alcohol abuse (as defined by an average daily consumption of alcohol > 30 g/day in men and > 20 g/day women), cirrhosis, autoimmune hepatitis and other causes of liver disease (viral hepatitis, hemochromatosis, Wilson's disease), drug induced hepatitis, chronic enteropathies, Chronic kidney disease

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Egyptian diabetic patients diagnosed with NAFLD
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
investigate adipokine dna polymorphism | 1 months
  to investigate adipokine gene polymorphism associated with prognosis of NAFLD patients
correlations | 1 month
  to correlate between gene polymorphism and glycated hemoglobin, liver enzyme and obesity

CONTACTS AND LOCATIONS:
Overall Officials: Amal Ahmed, PhD, Principal Investigator — professor
Locations (1):
- El Sahel teaching hospital, Cairo, Shobra, Egypt

IPD SHARING:
Plan to Share IPD: No